CLINICAL TRIAL: NCT00808015
Title: ASIA CHOICES CHampix Observational Investigation in the CEssation of Smoking
Brief Title: ASIA CHOICES CHampix (Varenicline) Observational Investigation in the CEssation of Smoking
Acronym: ASIA CHOICES
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: A3051112
Record Dates: First submitted 2008-12-12; First posted 2008-12-15 (Estimated); Results first posted 2011-07-28 (Estimated); Last update posted 2015-05-12 (Estimated); Status verified 2015-04

CONDITIONS: Smoking Cessation
Keywords: Observational non-interventional trial
MeSH Terms: conditions — Smoking Cessation | interventions — Varenicline

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients in routine practice: Patients prescribed Champix by treating physician and then entered into trial
  Interventions: Drug: varenicline

INTERVENTIONS:
Drug: varenicline — Champix will be prescribed as per usual practice and at the sole discretion of the physician
  Other Names: Champix, Chantix

SUMMARY:
The purpose of this study is to describe the characteristics of the smoker who wants to quit and his/her treating physician, in addition to determine the safety and effectiveness of Champix in the real-world setting of smokers in routine clinical practice.

DETAILED DESCRIPTION:
Sampling Method Description: Patients enrolled after being prescribed Champix for smoking cessation at the sole discretion of treating physician and patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients enrolled should meet the usual prescribing criteria for Champix® as per the local product information and should be entered into the trial at the investigator's discretion

Exclusion Criteria:

* All patients enrolled should meet the usual prescribing criteria for Champix® as per the local product information and should be entered into the trial at the investigator's discretion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study is in Asian patients. The patients enrolled should be of legal adult age who regularly smoke and whose main tobacco product is cigarettes. The patients must be willing to make an attempt to stop smoking.
Sampling Method: Non-Probability Sample
Enrollment: 1373 (Actual)
Dates: Start 2009-02; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (51):
- China (18):
  - Pfizer Investigational Site, Beijing, Beijing Municipality
  - Pfizer Investigational Site, Guangzhou, Guangdong
  - Pfizer Investigational Site, Shenzhen, Guangdong
  - Pfizer Investigational Site, Wuhan, Hubei
  - Pfizer Investigational Site, Changsha, Hunan
  - Pfizer Investigational Site, Nanjing, Jiangsu
  - Pfizer Investigational Site, Suzhou, Jiangsu
  - Pfizer Investigational Site, Shenyang, Liaoning
  - Pfizer Investigational Site, Xi'an, Shaanxi
  - Pfizer Investigational Site, Taiyuan, Shanxi
  - Pfizer Investigational Site, Chengdu, Sichuan
  - Pfizer Investigational Site, Tianjin, Tianjin Municipality
  - Pfizer Investigational Site, Beijing
  - Pfizer Investigational Site, Nanning
  - Pfizer Investigational Site, Shanghai
  - Pfizer Investigational Site, Shijiazhuang
  - Pfizer Investigational Site, Tianjin
  - Pfizer Investigational Site, Wuhan
- India (12):
  - Pfizer Investigational Site, Hyderabad, Andhra Pradesh
  - Pfizer Investigational Site, Ahmedabad, Gujarat
  - Pfizer Investigational Site, Kochi, Kerala
  - Pfizer Investigational Site, Tthiruvananthapuram, Kerala
  - Pfizer Investigational Site, Mumbai, Maharashtra
  - Pfizer Investigational Site, Delhi, National Capital Territory of Delhi
  - Pfizer Investigational Site, New Delhi, National Capital Territory of Delhi
  - Pfizer Investigational Site, Daryāganj, New Delhi
  - Pfizer Investigational Site, Delhi, New Delhi
  - Pfizer Investigational Site, New Delhi, New Delhi
  - Pfizer Investigational Site, Coimbatore, Tamil Nadu
  - Pfizer Investigational Site, Chennai
- Philippines (10):
  - Pfizer Investigational Site, San Juan City, Batangas
  - Pfizer Investigational Site, Batac, Ilocos Norte
  - Pfizer Investigational Site, San Fernando City, La Union
  - Pfizer Investigational Site, Angeles City, Pampanga
  - Pfizer Investigational Site, Urdaneta, Pangasinan
  - Pfizer Investigational Site, Tarlac City, Tarlac
  - Pfizer Investigational Site, Davao City
  - Pfizer Investigational Site, Marikina City
  - Pfizer Investigational Site, Pasay
  - Pfizer Investigational Site, Quezon City
- South Korea (11):
  - Pfizer Investigational Site, Cheonan-si, Chungcheongnam-do
  - Pfizer Investigational Site, Goyang-si, Gyeonggi-do
  - Pfizer Investigational Site, Seongnam-si, Gyeonggi-do
  - Pfizer Investigational Site, Suwon, Gyeonggi-do
  - Pfizer Investigational Site, Yangsan, Gyeongsangnam-do
  - Pfizer Investigational Site, Iksan-Si, Jeollabuk-do
  - Pfizer Investigational Site, Daegu
  - Pfizer Investigational Site, Daejeon
  - Pfizer Investigational Site, Incheon
  - Pfizer Investigational Site, Seoul
  - Pfizer Investigational Site, Suwon

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051112&StudyName=ASIA%20CHOICES%20CHampix%20Observational%20Investigation%20in%20the%20CEssation%20of%20Smoking

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 1429 participants were screened for this study and 1377 participants were assigned to the study treatment.
Groups:
- Varenicline: Varenicline 0.5 mg once daily orally from Day 1 and titrated up to 1 mg dose twice daily (BID) from Day 8 till Week 12 or Last Observed Study Visit.
Period: Overall Study
Arm/Group | Varenicline
Started | 1377
Treated | 1373
Completed | 1033
Not Completed | 344
Not completed — Death | 1
Not completed — Lack of Efficacy | 58
Not completed — Lost to Follow-up | 76
Not completed — Participants not willing to participate | 158
Not completed — Adverse Event | 22
Not completed — Other | 25
Not completed — Enrolled but not treated | 4

BASELINE CHARACTERISTICS:
Arm/Group | Varenicline
Number analyzed (Participants) | 1373
Age, Continuous [Mean (Standard Deviation); unit: Years] | 45.2 (12.5)
Sex/Gender, Customized [Number; unit: Participants]
  Male | 1279
  Female | 88
  Unspecified | 6
Smoking history: Total number of years participant smoked [Median (Full Range); unit: Years] — N = 1308 for the parameter analyzed.
  Years | 20.0 [1.0 to 70.0]
Smoking history: Average number of cigarettes smoked per day in the last year [Median (Full Range); unit: cigarettes] — N = 1299 for the parameter analyzed.
  cigarettes | 20.00 [1.00 to 90.00]
Smoking history: Longest period of abstinence in the last year [Median (Full Range); unit: Days] — N = 1269 for the parameter analyzed.
  Days | 0.0 [0.0 to 365.0]
Smoking history : Number of times the participant has attempted to quit in past year [Median (Full Range); unit: Quit attempts] — N = 1257 for the parameter analyzed. Scores were graded as none [(no attempt) to 3 or more attempts].
  Quit attempts | 0.0 [0.0 to 30.0]
Smoking history : Participant categorized based on number of attempt to quit in the past year [Number; unit: participants] — N = 1257 for the parameter analyzed.
  participants
    None | 738
    One | 285
    Two | 107
    Three or more | 127
Smoking history : Did participant live with someone who smoked [Number; unit: participants] — N = 1287 for the parameter analyzed.
  participants
    Yes | 247
    No | 1040
Smoking history : Did participant have frequent contact with someone who smoked [Number; unit: participants] — N = 1270 for the parameter analyzed.
  participants
    Yes | 1071
    No | 199
Smoking history: Lifetime serious quit attempts [Number; unit: participants] — A serious quit attempt was defined as smoking cessation for more than 24 hours. Scores were graded as none (no attempt) to 3 or more attempts). N = 649 for the parameter analyzed.
  participants
    None | 16
    One | 322
    Two | 117
    Three or more | 194
Quit History : Main reasons for relapses after previous attempts [Number; unit: participants] — N = 813 for the parameter analyzed.
  participants
    Family / Friends | 164
    Smoking is a habitual response to stress/pressure | 381
    Urge to smoke is too strong | 449
    Weight gain | 20
    Exposure to smoke environment | 227
Quit History : Reasons motivated participant to quit smoking [Number; unit: participants] — N = 1299 for the parameter analyzed.
  participants
    Health reasons | 1218
    Family / Friends | 902
    Money / cost | 72
    Body image / appearance | 78
    Smoking ban in public places | 37
Fagerstrom Test of Nicotine Dependence (FTND) [Mean (Standard Deviation); unit: Scores on a scale] — FTND was designed to provide measure of nicotine dependence related to cigarette smoking. It contains 4 yes-no and 2 multiple choice questions. Items are scored 0-3 for multiple choice items, items are summed to yield total score of 0-10 (0=minimum to 10=maximum nicotine dependence).N= 268 for the parameter analyzed.
  Scores on a scale | 5.50 (2.43)
Exhaled Carbon monoxide (CO) level [Mean (Standard Deviation); unit: parts per million (ppm)] — The CO level was measured from exhaled air of the participant using CO analyzer at the last observed study visit which was the last available CO level recorded after baseline. The CO level was only measured if it was a part of the usual practice at the site. N= 361 for the parameter analyzed.
  parts per million (ppm) | 14.20 (7.69)
Average number of cigarettes smoked per day in the previous 7 day period at baseline [Median (Full Range); unit: cigarettes] — The average number of cigarettes smoked per day over the last 7 days was collected as a part of nicotine use inventory assessment through consent record form module which included a questionnaire: Did the participant smoke any cigarettes (even a puff) in last 7 days (Yes/No) and Did the participant use any other tobacco products (example- pipe, cigars, chew, snuff) in last 7 days (Yes/No). N=1256 for the parameter analyzed.
  cigarettes | 20.0 [1.0 to 80.0]
Smoking related concurrent diseases [Number; unit: participants] — The 'n' is signifying those participants who were evaluated for this measure respectively.
  participants
    Occlusive disease of non-coronary arteries(n=1183) | 21
    Atherosclerotic vascular disease (n=1181) | 138
Cardiovascular risk factors [Number; unit: participants] — N=138 for the parameter analyzed.
  participants
    Family history of Cardiovascular disease or stroke | 111
    Left ventricular hypertrophy | 13
    Unspecified | 13
    History of microalbuminuria | 9
    Documented Ankle Brachial Index (ABI) <0.9 | 3
Participant social status : Current Marital Status [Number; unit: participants] — N = 1258 for the parameter analyzed.
  participants
    Married | 1124
    Never Married | 104
    Divorced | 13
    Widowed | 12
    Separated | 4
    Cohabitating | 1
Participant social status : Current Living Situation [Number; unit: participants] — N = 1243 for the parameter analyzed.
  participants
    Living with a spouse or significant other | 1002
    Living with other family member(s) or roommate(s) | 193
    Living alone | 45
    Living in residential treatment center | 1
    Living in institution | 1
    Other unspecified | 1
Healthcare utilization status: Reimbursement type [Number; unit: participants] — N=1287 for the parameter analyzed.
  participants
    Private Insurance | 111
    No Insurance | 276
    Public Insurance | 877
    Other unspecified | 23
Health care utilization: Employment status [Number; unit: participants] — N=1266 for the parameter analyzed.
  participants
    Not employed | 235
    Full-time employed | 1016
    Part-time employed | 15
Family history of mental illness [Number; unit: participants] — Family members who were considered for the following parameter were Biological Parents, Biological Siblings, Children and Grandparents. The 'n' is signifying those participants who were evaluated for this measure respectively.
  participants
    Alcohol abuse (n=122) | 12
    Cerebral apoplexy (n=1) | 1
    Dementia (n=120) | 2
    Depression (Chronic or recurrent) (n=119) | 2
    Dissociative disorder (n=1) | 1
    Major depression (n=120) | 1
    Mental disorder (n=1) | 1
    Nicotine addiction (n=8) | 8
    Parkinson's disease (n=1) | 1
    Schizophrenia (n=120) | 4
Nondrug treatments / procedures for primary diagnosis [Number; unit: participants] — N=701 for the parameter analyzed.
  participants
    Smoking Cessation Counseling | 661
    Quit Smoking Clinic | 190
    Other unspecified | 1
Prior Drug Treatment [Number; unit: participants] — N=435 for the parameter analyzed.
  participants
    Acamprosate | 2
    Acarbose | 14
    Aceclofenac | 1
    Acetylcarnitine | 1
    Acetylcysteine | 11
    Acetylsalicylic acid | 99
    Acetylsalicylic acid/atorvastatin/ramipril | 1
    Acetylsalicylic acid/clopidogrel | 1
    Adenine/biphenyldimethyldicarboxylate/vitamins | 1
    Alfuzosin | 1
    All other therapeutic products | 6
    Allopurinol | 2
    Almagate | 4
    Alprazolam | 6
    Ambroxol | 4
    Ambroxol acefyllinate | 1
    Ambroxol hydrochloride | 8
    Aminophylline | 2
    Amisulpride | 1
    Amitriptyline hydrochloride | 2
    Amlodipine | 17
    Amlodipine besilate | 17
    Amlodipine besilate/atorvastatin calcium | 2
    Amlodipine besylate/valsartan | 2
    Amlodipine camsilate | 2
    Amlodipine maleate | 2
    Amlodipine orotate | 2
    Amlodipine/valsartan | 3
    Amoxicillin | 6
    Amoxicillin sodium | 1
    Antisterone | 2
    Aripiprazole | 1
    Aronamin gold | 1
    Arotinolol hydrochloride | 1
    Artemisia asiatica | 1
    Artemisia asiatica/ethanol | 1
    Asmeton | 9
    Atenolol | 2
    Atorvastatin | 44
    Atorvastatin calcium | 9
    Azathioprine | 2
    Azelastine | 2
    Azelastine hydrochloride | 2
    Azithromycin | 3
    Aztreonam | 1
    B-komplex "leciva" | 1
    Bambuterol hydrochloride | 1
    Becosules syrup | 2
    Becosym forte | 1
    Becotal | 1
    Benazepril | 1
    Benazepril hydrochloride | 2
    Benproperine | 1
    Benproperine phosphate | 1
    Bepotastine besilate | 2
    Beraprost | 1
    Betahistine | 1
    Bevantolol | 1
    Biphenyl dimethyl dicarboxylate/garlic | 1
    Biselect | 1
    Bismuth subcitrate tripotassium | 1
    Bismuth subcitrate tripotassium/ranitidine HCl | 2
    Bisoprolol | 6
    Bisoprolol fumarate | 12
    Borneol/notoginseng/salvia miltiorrhiza | 1
    Bromelains/dehydrocholic/pancreatin/simeticone | 1
    Broncho-vaxom | 2
    Budesonide | 2
    Bupropion | 1
    Bupropion hydrochloride | 1
    Buspiron | 1
    Buspirone | 1
    Calcium chloride | 1
    Calcium citrate/colecalciferol | 1
    Calcium lactate | 1
    Candesartan | 6
    Candesartan cilexetil | 2
    Carbazochrome | 1
    Cardiovascular system drugs | 1
    Carvedilol | 7
    Cefaclor | 5
    Cefoperazone sodium | 2
    Cefpodoxime | 1
    Cefpodoxime proxetil | 1
    Cefradine | 1
    Ceftriaxone sodium | 1
    Cefuroxime | 3
    Cefuroxime sodium | 1
    Cephalosporins and related substances | 2
    Cetirizine | 1
    Chlormadinone acetate | 1
    Choline alfoscerate | 5
    Chondroitin/glucosamine | 1
    Cilazapril | 2
    Cilnidipine | 6
    Cilostazol | 3
    Cimetidine | 1
    Ciprofloxacin | 2
    Citalopram | 1
    Clarithromycin | 5
    Clobazam | 1
    Clonazepam | 3
    Clopidogrel | 19
    Clopidogrel sulfate | 16
    Co-diovan | 2
    Colchicine | 2
    Cordalin /old form | 1
    Cough syrup | 1
    Dexamethasone | 1
    Dexamethasone/neomycin sulfate/polymyxin B sulfate | 1
    Diacerein | 1
    Diazepam | 2
    Diclofenac | 1
    Digoxin | 2
    Dihydrocodeine bitartrate | 2
    Diltiazem | 6
    Diltiazem hydrochloride | 1
    Dimenhydrinate | 1
    Diprophylline | 1
    Disulfiram | 1
    Domperidone | 4
    Donepezil | 1
    Doxazosin mesilate | 1
    Doxofylline | 14
    Drug, unspecified | 3
    Duloxetine hydrochloride | 1
    Ecabet monosodium | 1
    Efavirenz/emtricitabine/tenofovir | 1
    Efonidipine | 1
    Enalapril | 2
    Enalapril maleate | 1
    Enzymes | 1
    Epoprostenol | 1
    Eprosartan | 2
    Eprosartan mesilate | 1
    Eprosartan mesilate/hydrochlorothiazide | 2
    Erdosteine | 6
    Ergenyl chrono | 2
    Erlotinib hydrochloride | 1
    Erythromycin ethylsuccinate | 1
    Escitalopram | 3
    Esomeprazole | 3
    Esomeprazole magnesium | 3
    Etizolam | 1
    Etoposide | 1
    Etoricoxib | 1
    Ezetimibe | 1
    Ezetimibe/simvastatin | 4
    Famotidine | 2
    Felodipine | 7
    Fenofibrate | 10
    Ferric hydroxide polymaltose complex | 1
    Ferrous sulfate | 1
    Fexofenadine | 1
    Fish oil | 1
    Flumazenil | 1
    Flunarizine | 1
    Fluoxetine | 2
    Folic acid | 4
    Formoterol | 3
    Formoterol fumarate | 2
    Fosinopril | 3
    Fosinopril sodium | 2
    Furosemide | 2
    Gabapentin | 1
    Gefarnate | 1
    General nutrients/herbal NOS | 1
    Ginkgo biloba | 1
    Glibenclamide | 1
    Gliclazide | 10
    Glimepiride | 12
    Glimepiride/metformin hydrochloride | 1
    Glipizide | 3
    Gliquidone | 1
    Glucose | 2
    Glyceryl trinitrate | 4
    Guaifenesin | 1
    Hedera helix | 4
    Herbal preparation | 13
    Homeopatic preparation | 8
    Hyaluronate sodium | 1
    Hydrochlorothiazide | 7
    Hydrocortisone | 1
    Hydrotalcite | 1
    Hyzaar | 2
    Indapamide | 1
    Indometacin | 1
    Infliximab | 1
    Inosine | 1
    Insulin | 8
    Insulin aspart | 1
    Insulin glargine | 2
    Insulin glulisine | 1
    Insulin human | 3
    Insulin human injection, isophane | 2
    Ipratropium | 1
    Ipratropium bromide | 4
    Irbesartan | 13
    Isosorbide dinitrate | 2
    Isosorbide mononitrate | 11
    Isotretinoin | 1
    Itavastatin | 6
    Itopride | 1
    Itopride hydrochloride | 1
    Karvea hct | 3
    Kombipak II | 1
    Lacidipine | 1
    Lactitol | 1
    Lamivudine | 3
    Lansoprazole | 1
    Lekovit Ca | 2
    Lercanidipine | 1
    Lercanidipine hydrochloride | 1
    Levamlodipine besylate | 2
    Levocloperastine fendizoate | 3
    Levodropropizine | 4
    Levofloxacin | 8
    Levofloxacin hydrochloride | 5
    Levosalbutamol hydrochloride | 1
    Levosulpiride | 3
    Levothyroxine sodium | 3
    Liquorice | 1
    Lisinopril | 2
    Lithium carbonate | 1
    Loratadine | 1
    Lorazepam | 1
    Losartan | 7
    Losartan potassium | 8
    Magnesium hydroxide | 2
    Mecobalamin | 1
    Medilac-S | 1
    Mesalazine | 1
    Metformin | 29
    Metformin hydrochloride | 15
    Metformin hydrochloride/rosiglitazone | 1
    Metformin hydrochloride/sitagliptin | 1
    Methoxyphenamine | 1
    Methylprednisolone | 3
    Metoprolol | 11
    Metoprolol succinate | 3
    Metoprolol tartrate | 6
    Midazolam | 2
    Milnacipran hydrochloride | 1
    Mirtazapine | 1
    Molsidomine | 2
    Mometasone | 1
    Montelukast | 3
    Montelukast sodium | 4
    Mosapride | 1
    Mosapride citrate | 4
    Moxifloxacin hydrochloride | 2
    Multivitamins, plain | 2
    Myrtol | 3
    Naltrexone | 1
    Nateglinide | 4
    Nebivolol | 1
    Nicorandil | 5
    Nicotinic acid | 2
    Nifedipine | 16
    Nimodipine | 2
    Nisoldipine | 1
    Nitrendipine | 1
    Olanzapine | 2
    Olmesartan | 5
    Omega-3 marine triglycerides | 1
    Omega-3 triglycerides | 3
    Omeprazole | 3
    Orlistat | 2
    Oxazepam | 2
    Oxcarbazepine | 1
    Oxycodone hydrochloride | 1
    Pantoprazole | 1
    Pantoprazole sodium | 4
    Paracetamol | 5
    Paroxetine | 1
    Paroxetine hydrochloride | 1
    Penicillin NOS | 1
    Perindopril | 8
    Pethidine hydrochloride | 1
    Phenytoin sodium | 1
    Phosphatidyl choline | 1
    Pioglitazone | 3
    Pioglitazone hydrochloride | 3
    Pip/tazo | 1
    Platelets, human blood | 1
    Polycarbophil calcium | 1
    Pranlukast hydrate | 1
    Pravastatin | 7
    Pravastatin sodium | 4
    Prednisolone | 4
    Pregabalin | 2
    Procaterol | 2
    Propranolol | 1
    Propranolol hydrochloride | 1
    Pseudoephedrine hydrochloride | 1
    Pyridoxine hydrochloride | 1
    Quetiapine fumarate | 2
    Rabeprazole | 3
    Rabeprazole sodium | 2
    Ramipril | 4
    Ranitidine | 1
    Ranitidine hydrochloride | 3
    Rebamipide | 12
    Repaglinide | 3
    Risedronic acid | 1
    Risperidone | 2
    Rosiglitazone maleate | 1
    Rosuvastatin | 14
    Rosuvastatin calcium | 1
    Roxithromycin | 1
    Salbutamol | 7
    Salbutamol sulfate | 1
    Salmeterol | 1
    Salmeterol xinafoate | 3
    Salvia miltiorrhiza | 1
    Sarpogrelate hydrochloride | 2
    Selective beta-2-adrenoreceptor agonists | 1
    Selegiline hydrochloride | 1
    Seretide mite | 15
    Sertraline | 1
    Sibutramine | 1
    Sildenafil citrate | 2
    Silymarin | 1
    Simvastatin | 19
    Sinemet | 1
    Sinilgel | 1
    Sitagliptin | 6
    Sodium chloride | 1
    Sotalol hydrochloride | 1
    Spironolactone | 2
    Streptomycin | 1
    Sucralfate | 1
    Sulglicotide | 2
    Sulodexide | 1
    Symbicort turbuhaler "draco" | 6
    Tamsulosin | 5
    Tamsulosin hydrochloride | 3
    Tazobactam sodium | 2
    Telmisartan | 8
    Terazosin | 1
    Terazosin hydrochloride | 1
    Terbutaline sulfate | 1
    Theophylline | 7
    Thiamazole | 2
    Thioctic acid | 1
    Throat preparations | 1
    Tianeptine | 1
    Ticlopidine | 1
    Tiotropium | 10
    Tiotropium bromide | 2
    Tiotropium bromide/formoterol fumarate | 1
    Tiropramide hydrochloride | 2
    Tocopherol | 1
    Tramadol hydrochloride | 1
    Tranexamic acid | 3
    Travad phosphate enema | 1
    Trazodone | 1
    Triaprin | 1
    Triflusal | 1
    Trimetazidine | 2
    Trimetazidine hydrochloride | 2
    Udenafil | 1
    Ultracet | 3
    Ursodeoxycholic acid | 4
    Valproate semisodium | 1
    Valsartan | 9
    Verapamil | 1
    Vildagliptin | 1
    Vitamins | 1
    Vitamins with minerals | 1
    Voglibose | 3
    Warfarin | 6
    Yeast | 1
    Zevit | 1
    Zolpidem | 5
    Zolpidem tartrate | 3
Medical History [Number; unit: participants] — N=129 for the parameter analyzed.
  participants
    Acute myocardial infarction | 2
    Angina pectoris | 18
    Arrhythmia | 3
    Arteriosclerosis coronary artery | 1
    Atrial fibrillation | 5
    Bundle branch block right | 1
    Cardiac failure | 1
    Cardiac failure congestive | 2
    Cardiac valve disease | 1
    Congestive cardiomyopathy | 1
    Cor pulmonale chronic | 1
    Coronary artery disease | 72
    Coronary artery stenosis | 1
    Left ventricular hypertrophy | 1
    Mitral valve calcification | 1
    Myocardial infarction | 1
    Myocardial ischaemia | 1
    Prinzmetal angina | 2
    Sinus tachycardia | 1
    Ventricular extrasystoles | 1
    Hearing impaired | 1
    Basedow's disease | 2
    Goitre | 1
    Hyperthyroidism | 3
    Hypothyroidism | 5
    Thyroid cyst | 1
    Blindness unilateral | 1
    Visual impairment | 1
    Abdominal discomfort | 1
    Abdominal pain upper | 1
    Colitis | 1
    Colonic polyp | 3
    Constipation | 3
    Crohn's disease | 1
    Diverticulum intestinal | 1
    Duodenal ulcer | 6
    Duodenitis | 1
    Dyspepsia | 5
    Gastric haemorrhage | 1
    Gastric ulcer | 6
    Gastritis | 53
    Gastritis atrophic | 4
    Gastritis erosive | 4
    Gastrooesophageal reflux disease | 11
    Haemorrhoids | 1
    Intestinal polyp | 1
    Irritable bowel syndrome | 2
    Nausea | 1
    Oesophagitis | 2
    Pancreatitis | 2
    Pancreatitis chronic | 1
    Peptic ulcer | 50
    Periodontitis | 1
    Reflux oesophagitis | 11
    Chest pain | 2
    Fatigue | 3
    Malaise | 1
    Pain | 1
    Alcoholic liver disease | 1
    Cholecystitis | 2
    Cholelithiasis | 1
    Chronic hepatitis | 2
    Hepatic cyst | 1
    Hepatic steatosis | 12
    Hepatitis | 2
    Hepatitis alcoholic | 1
    Behcet's syndrome | 1
    Sarcoidosis | 1
    Appendicitis | 1
    Body tinea | 1
    Bronchiectasis | 5
    Bronchitis | 15
    Chronic sinusitis | 1
    Cystitis | 1
    Helicobacter infection | 1
    Hepatitis B | 3
    Lower respiratory tract infection | 1
    Lung abscess | 1
    Nasopharyngitis | 1
    Onychomycosis | 1
    Pharyngitis | 12
    Pneumonia | 7
    Pulmonary tuberculosis | 8
    Pyelonephritis acute | 1
    Rhinitis | 7
    Tinea pedis | 2
    Tonsillitis | 1
    Tuberculosis | 3
    Tuberculosis gastrointestinal | 1
    Tuberculous pleurisy | 2
    Upper respiratory tract infection | 2
    Meniscus lesion | 1
    Blood cholesterol increased | 1
    Blood viscosity increased | 1
    HIV test positive | 1
    Hepatitis B virus test | 1
    Liver function test abnormal | 1
    Calcium deficiency | 1
    Diabetes mellitus | 132
    Dyslipidaemia | 167
    Gout | 1
    Hypercholesterolaemia | 2
    Hyperhomocysteinaemia | 1
    Hyperlipidaemia | 19
    Hyperuricaemia | 5
    Impaired fasting glucose | 1
    Iron deficiency | 1
    Obesity | 7
    Ankylosing spondylitis | 1
    Arthritis | 1
    Back pain | 1
    Intervertebral disc disorder | 1
    Neck pain | 1
    Osteoarthritis | 2
    Osteopenia | 1
    Osteoporosis | 4
    Rheumatoid arthritis | 4
    Acute lymphocytic leukaemia | 1
    Benign lung neoplasm | 1
    Brain neoplasm | 1
    Cervix carcinoma | 1
    Extranodal marginal zone B-cell lymphoma | 1
    Gastric adenoma | 1
    Gastric cancer | 1
    Head and neck cancer | 2
    Hepatic neoplasm malignant | 1
    Histiocytosis haematophagic | 1
    Laryngeal cancer | 1
    Leiomyosarcoma | 1
    Lung neoplasm | 9
    Lung neoplasm malignant | 8
    Prostate cancer | 1
    Rectal cancer | 2
    Renal cancer | 2
    Renal cell carcinoma | 1
    Renal neoplasm | 1
    Carotid artery occlusion | 1
    Carotid artery stenosis | 3
    Cerebral arteriosclerosis | 1
    Cerebral infarction | 4
    Cerebral ischaemia | 1
    Cerebrovascular accident | 21
    Dementia | 1
    Dizziness | 2
    Headache | 6
    Myasthenia gravis | 1
    Neuropathy peripheral | 1
    Parkinson's disease | 1
    Sedation | 1
    Transient ischaemic attack | 2
    Alcohol abuse | 46
    Bipolar disorder | 2
    Depressed mood | 1
    Depression | 8
    Dysthymic disorder | 1
    Generalised anxiety disorder | 11
    Insomnia | 5
    Major depression | 17
    Obsessive-compulsive disorder | 1
    Panic attack | 5
    Panic disorder | 6
    Personality disorder | 5
    Psychotic disorder | 1
    Schizoaffective disorder | 1
    Schizophrenia | 3
    Sleep disorder | 4
    Social phobia | 2
    Substance abuse | 14
    Bladder irritation | 1
    Nephrolithiasis | 1
    Proteinuria | 1
    Renal failure chronic | 2
    Benign prostatic hyperplasia | 9
    Erectile dysfunction | 2
    Organic erectile dysfunction | 1
    Asthma | 65
    Bronchitis chronic | 19
    Chronic obstructive pulmonary disease | 116
    Cough | 6
    Dyspnoea | 3
    Emphysema | 7
    Epistaxis | 1
    Haemoptysis | 3
    Idiopathic pulmonary fibrosis | 1
    Interstitial lung disease | 3
    Pleural effusion | 1
    Pneumothorax | 1
    Pulmonary bulla | 1
    Pulmonary embolism | 1
    Pulmonary mass | 3
    Respiratory disorder | 2
    Rhinitis allergic | 7
    Sleep apnoea syndrome | 5
    Snoring | 1
    Acne | 1
    Alopecia areata | 1
    Dermatitis contact | 1
    Pruritus | 1
    Urticaria | 1
    Alcoholic | 1
    Aortic valve replacement | 1
    Haemorrhoid operation | 1
    Arteriosclerosis | 2
    Hypertension | 229
    Peripheral vascular disorder | 2
    Thromboangiitis obliterans | 2
    Vasculitis | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Smoking Abstinence at Week 12
Description: Four criteria used for derivation of smoking abstinence status: if participant smoked any cigarettes (even a puff) in last 7 days (Yes/No); if participant used any other tobacco products in last 7 days (Yes/No); average number of cigarettes smoked per day over last 7 days (in cigarettes/day); CO level (positive: if more than 10 ppm; negative : if 0-10 ppm).Smoking abstinence status was determined as: smoking: if participant responded positively to at least 1 of above 4; quit: if participant responded negatively to all 4; unknown: if participant had missing information for all 4.
Time Frame: Week 12
Population: Full analysis set (FAS) included all participants who received at least 1 dose of study medication
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 1373
percentage of participants | 46.40 [43.73 to 49.07]

2. Secondary Outcome: Percentage of Participants With Smoking Abstinence Before Last Observed Study Visit
Description: as for outcome 1
Time Frame: Last observed study visit (Week 12 or early termination [ET])
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 1373
percentage of participants | 50.30 [47.58 to 52.93]

3. Secondary Outcome: Percentage of Participants With Smoking Abstinence Status From Week 3 to Week 11
Description: as for outcome 1
Time Frame: Week 3 through Week 11
Population: At Week t (t = 3 to 11), the analysis population was "Observed Cases minus Week t" (OC minus Week t), that is (i-e), participants in FAS excluding missing values at the time point in question where OC was the subset of participants in FAS with observed (not missing) values.
Measure: Number; unit: percentage of participants
Arm/Group | Varenicline
Number analyzed (Participants) | 1373
percentage of participants
  Week 3 (n= 677) | 31.3
  Week 4 (n= 799) | 38.2
  Week 5 (n= 988) | 45.4
  Week 6 (n= 959) | 47.8
  Week 7 (n= 888) | 49.5
  Week 8 (n= 812) | 51.6
  Week 9 (n= 765) | 55.2
  Week 10 (n= 702) | 55.4
  Week 11 (n= 605) | 59.2

4. Secondary Outcome: CO Level at Last Observed Study Visit
Description: The CO level was measured from exhaled air of the participant using CO analyzer at the last observed study visit which was the last available CO level recorded after baseline. The CO level was only measured if it was a part of the usual practice at the site.
Time Frame: Last observed study visit (Week 12 or ET)
Population: FAS population included all participants who received at least 1 dose of study medication during study. Missing observations were not imputed and hence the participants analyzed were those without missing values (N=115).
Measure: Mean (Standard Deviation); unit: ppm
Arm/Group | Varenicline
Number analyzed (Participants) | 115
ppm | 4.1 (4.81)

5. Secondary Outcome: Average Weekly Number of Cigarettes Smoked at Last Observed Study Visit
Description: The average number of cigarettes smoked per day over the last 7 days was collected as a part of nicotine use inventory assessment through consent record form module which included a questionnaire: Did the participant smoke any cigarettes (even a puff) in last 7 days (Yes/No) and Did the participant use any other tobacco products (example- pipe, cigars, chew, snuff) in last 7 days (Yes/No).
Time Frame: Last observed study visit (Week 12 or ET)
Population: FAS population included all participants who received at least 1 dose of study medication during study. Missing observations were not imputed and hence the participants analyzed were those without missing values (N=518).
Measure: Median (Full Range); unit: cigarettes
Arm/Group | Varenicline
Number analyzed (Participants) | 518
cigarettes | 10.0 (9.57) [1.0 to 80.0]

6. Other Pre Specified Outcome: Varenicline Prescription Status
Description: Prescribed status was assessed using the following question in consent record form: Would a maintenance period of the drug be prescribed to the participant after this study ends (Yes/No). Missing values were recorded as 'unknown'.
Time Frame: After last observed study visit (Week 12 or ET)
Population: FAS population included all participants who received at least 1 dose of study medication.
Measure: Number; unit: participants
Arm/Group | Varenicline
Number analyzed (Participants) | 1373
participants
  Prescription status = Yes | 145
  Prescription status = No | 962
  Prescription status = Unknown | 266

7. Other Pre Specified Outcome: Average Daily Dose of Varenicline
Time Frame: Days 1-3, Days 4-7, Day 8 through last observed study visit (Week 12 or ET)
Population: FAS population included all participants who received at least 1 dose of study treatment. Missing values were excluded from analysis. The 'n' is signifying those participants who received study drug and were evaluated for this measure at the timepoint for each group respectively.
Measure: Median (Full Range); unit: mg
Arm/Group | Varenicline
Number analyzed (Participants) | 1373
mg
  Days 1-3 | 0.5 (0.13) [0.5 to 2.0]
  Days 4-7 (n=1347) | 1.0 (0.21) [0.5 to 2.0]
  Day 8 - Last observed study visit (n=1284) | 2.0 (0.27) [0.5 to 2.0]

8. Other Pre Specified Outcome: Median Duration of Treatment of Varenicline
Description: The duration was defined as the total number of dosing days from first to last day of each study treatment.
Time Frame: Baseline through last observed study visit (Week 12 or ET)
Population: FAS population included all participants who received at least 1 dose of study treatment. Missing values were excluded from analysis.
Measure: Median (Full Range); unit: Days
Arm/Group | Varenicline
Number analyzed (Participants) | 1373
Days | 43.0 [1.0 to 271.0]

9. Other Pre Specified Outcome: Concomitant Drug Treatments
Time Frame: Baseline through Last observed study visit (Week 12 or ET)
Population: FAS included all participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Varenicline
Number analyzed (Participants) | 1373
Participants
  Acamprosate | 5
  Acarbose | 17
  Aceclofenac | 1
  Acetylcarnitine | 2
  Acetylcysteine | 14
  Acetylsalicylic acid | 110
  Acetylsalicylic acid/atorvastatin/ramipril | 1
  Acetylsalicylic acid/clopidogrel | 1
  Adenine/biphenyldimethyldicarboxylate/vitamins | 1
  Albumin human | 1
  Alfuzosin | 1
  All other therapeutic products | 11
  Allopurinol | 2
  Almagate | 8
  Almagel | 1
  Alprazolam | 8
  Aluminum hydroxide/magnesium carbonate | 1
  Amantadine hydrochloride / paracetamol | 1
  Ambroxol | 3
  Ambroxol acefyllinate | 3
  Ambroxol hydrochloride | 4
  Amikacin | 1
  Amino acids | 2
  Amino acids NOS/carbohydrates NOS/electrolytes NOS | 1
  Aminophylline | 1
  Amisulpride | 2
  Amitriptyline hydrochloride | 2
  Amlodipine | 18
  Amlodipine besilate | 21
  Amlodipine besilate/atorvastatin calcium | 3
  Amlodipine besilate/valsartan | 2
  Amlodipine camsilate | 2
  Amlodipine maleate | 2
  Amlodipine orotate | 2
  Amlodipine/valsartan | 3
  Ammonium Cl/chlorpheniramine maleate | 1
  Amoxicillin | 1
  Amoxicillin sodium | 1
  Anisodamine | 1
  Antacids | 1
  Antidiarrhoeal microorganisms | 1
  Antisterone | 2
  Aripiprazole | 1
  Aronamin gold | 1
  Arotinolol hydrochloride | 1
  Artemisia asiatica | 1
  Artemisia asiatica/ethanol | 1
  Asasantin | 1
  Asmeton | 8
  Atenolol | 4
  Atorvastatin | 54
  Atorvastatin calcium | 7
  Atorvastatin/fenofibrate | 2
  Azathioprine | 2
  Azelastine | 2
  Azelastine hydrochloride | 5
  Azithromycin | 6
  Aztreonam | 1
  B-komplex "leciva" | 1
  Bambuterol hydrochloride | 1
  Becosules syrup | 2
  Becosym forte | 1
  Becotal | 1
  Benazepril | 1
  Benazepril hydrochloride | 2
  Benexate hydrochloride | 1
  Benproperine | 1
  Benproperine phosphate | 3
  Benzodiazepine derivatives | 1
  Bepotastine besilate | 2
  Beraprost | 1
  Beraprost sodium | 1
  Berberine | 1
  Beszyme | 1
  Betahistine | 1
  Bevantolol | 1
  Biselect | 1
  Bismuth subcitrate tripotassium | 1
  Bismuth subcitrate tripotassium/ranitidine HCl | 2
  Bisoprolol | 6
  Bisoprolol fumarate | 13
  Borneol/notoginseng/salvia miltiorrhiza | 1
  Bromelains/dehydrocholic/pancreatin/simeticone | 1
  Bromhexine | 3
  Broncho-vaxom | 2
  Budesonide | 4
  Bufferin | 1
  Bupropion | 3
  Bupropion hydrochloride | 1
  Buspiron | 1
  Buspirone | 1
  Calcitriol / calcium citrate | 1
  Calcium citrate/colecalciferol | 1
  Calcium lactate | 1
  Candesartan | 7
  Candesartan cilexetil | 2
  Carbazochrome | 1
  Cardiovascular system drugs | 1
  Carvedilol | 7
  Cefaclor | 3
  Cefalexin | 1
  Cefcapene pivoxil hydrochloride | 2
  Cefixime | 5
  Cefoperazone sodium | 1
  Cefpodoxime | 3
  Cefpodoxime proxetil | 1
  Cefradine | 1
  Ceftriaxone | 1
  Ceftriaxone sodium | 2
  Cefuroxime | 1
  Cefuroxime axetil | 1
  Cefuroxime sodium | 3
  Celecoxib | 1
  Cephalosporins and related substances | 2
  Cetirizine | 1
  Chlordiazepoxide/clidinium bromide/dicycloverine | 4
  Chlormadinone acetate | 1
  Chlorphenamine maleate | 2
  Chlorphenesin carbamate | 1
  Choline alfoscerate | 7
  Chondroitin/glucosamine | 1
  Cilazapril | 2
  Cilnidipine | 7
  Cilostazol | 5
  Cimetidine | 3
  Cimetropium bromide | 1
  Cinnarizine | 1
  Ciprofloxacin | 2
  Ciprofloxacin hydrochloride | 1
  Citalopram | 1
  Citicoline | 1
  Clarithromycin | 4
  Clavulin | 2
  Clobazam | 1
  Clonazepam | 7
  Clopidogrel | 21
  Clopidogrel sulfate | 16
  Co-diovan | 2
  Colchicine | 3
  Cordalin/old form/ | 1
  Cotylenol | 1
  Cough syrup | 1
  Cyproterone acetate | 1
  Desmopressin | 1
  Desonide | 1
  Dexamethasone | 3
  Dexamethasone/neomycin sulfate/polymyxin B sulfate | 1
  Diazepam | 4
  Diclofenac | 1
  Digoxin | 3
  Dihydrocodeine bitartrate | 3
  Diloxanide furoate/metronidazole | 1
  Diltiazem | 6
  Diltiazem hydrochloride | 1
  Dimenhydrinate | 1
  Disulfiram | 1
  Docetaxel | 1
  Domperidone | 7
  Domperidone maleate | 1
  Domperidone/pantoprazole | 2
  Domperidone/rabeprazole | 1
  Domperidone/rabeprazole sodium | 1
  Donepezil | 1
  Doxazosin | 1
  Doxazosin mesilate | 1
  Doxofylline | 21
  Drotaverine | 1
  Drug, unspecified | 5
  Duloxetine | 1
  Duloxetine hydrochloride | 1
  Ebastine | 2
  Ecabet monosodium | 3
  Efavirenz/emtricitabine/tenofovir | 1
  Efonidipine | 1
  Enalapril | 3
  Enalapril maleate | 1
  Epoprostenol | 1
  Eprosartan | 2
  Eprosartan mesilate | 1
  Eprosartan mesilate/hydrochlorothiazide | 2
  Erdosteine | 14
  Ergenyl chrono | 3
  Erlotinib hydrochloride | 1
  Erythromycin ethylsuccinate | 1
  Escitalopram | 3
  Esomeprazole | 2
  Esomeprazole magnesium | 2
  Estazolam | 1
  Etizolam | 2
  Etoposide | 1
  Etoricoxib | 1
  Ezetimibe | 1
  Ezetimibe/simvastatin | 4
  Famotidine | 2
  Felodipine | 7
  Fenofibrate | 11
  Ferric hydroxide polymaltose complex | 1
  Ferrous sulfate | 1
  Fexofenadine | 3
  Fexofenadine hydrochloride | 1
  Fish oil | 1
  Flunarizine | 1
  Fluoxetine | 4
  Fluoxetine hydrochloride | 1
  Fluticasone propionate | 1
  Fluvastatin | 1
  Folic acid | 4
  Folic acid/mecobalamin/pyridoxine hydrochloride | 2
  Foraseq | 1
  Formoterol | 3
  Formoterol fumarate | 1
  Fosinopril | 3
  Fosinopril sodium | 2
  Furosemide | 3
  Gabapentin | 2
  Galenic /fluticasone/salmeterol | 2
  Galenic /salbutamol/guaifenesin | 1
  General nutrients/minerals/vitamins | 1
  Ginkgo biloba | 1
  Ginkgo biloba extract | 1
  Glibenclamide | 1
  Gliclazide | 12
  Glimepiride | 13
  Glimepiride/metformin | 2
  Glimepiride/metformin hydrochloride | 2
  Glipizide | 3
  Gliquidone | 1
  Glucose | 2
  Glyceryl trinitrate | 4
  Guaifenesin | 1
  Hedera helix | 6
  Heparin-fraction | 1
  Hepatitis B vaccine | 1
  Herbal preparation | 13
  Homeopatic preparation | 9
  Hyaluronate sodium | 2
  Hydrochlorothiazide | 8
  Hydrotalcite | 3
  Hydroxychloroquine | 1
  Hydroxyzine | 1
  Hydroxyzine hydrochloride | 1
  Hyoscine butylbromide | 2
  Hyzaar | 2
  I.v. solutions | 2
  Ibuprofen | 2
  Indapamide | 2
  Indometacin | 1
  Infliximab | 1
  Inosine | 1
  Insulin | 10
  Insulin aspart | 1
  Insulin glargine | 2
  Insulin glulisine | 1
  Insulin human | 3
  Insulin human injection, isophane | 2
  Ipratropium | 1
  Ipratropium bromide | 4
  Irbesartan | 14
  Isoconazole nitrate | 1
  Isosorbide dinitrate | 3
  Isosorbide mononitrate | 11
  Isotretinoin | 1
  Ispaghula | 1
  Ispaghula husk | 1
  Itavastatin | 8
  Itopride | 1
  Itopride hydrochloride | 1
  Itraconazole | 3
  Karvea hct | 3
  Kombipak II | 1
  Lacidipine | 1
  Lactitol | 1
  Lactulose | 3
  Lamivudine | 3
  Lansoprazole | 3
  Lekovit Ca | 2
  Lenograstim | 1
  Lercanidipine | 1
  Lercanidipine hydrochloride | 1
  Levamlodipine besylate | 2
  Levocarnitine | 3
  Levocetirizine | 1
  Levocetirizine dihydrochloride | 1
  Levocetirizine dihydrochloride/montelukast sodium | 1
  Levocloperastine fendizoate | 2
  Levodropropizine | 3
  Levofloxacin | 14
  Levofloxacin hydrochloride | 2
  Levosalbutamol hydrochloride | 1
  Levosulpiride | 6
  Levothyroxine sodium | 4
  Lipase | 1
  Lisinopril | 2
  Lithium carbonate | 1
  Loperamide | 1
  Loratadine | 2
  Lorazepam | 3
  Losartan | 9
  Losartan potassium | 10
  Magnesium hydroxide | 3
  Magnesium oxide | 2
  Mecobalamin | 4
  Medilac-S | 3
  Mefloquine | 1
  Megestrol acetate | 1
  Meprobamate | 1
  Meropenem | 1
  Mesalazine | 2
  Metformin | 32
  Metformin hydrochloride | 16
  Metformin hydrochloride/rosiglitazone | 1
  Metformin hydrochloride/sitagliptin | 1
  Methoxyphenamine | 1
  Methylprednisolone | 6
  Metoclopramide | 2
  Metoclopramide hydrochloride | 2
  Metoprolol | 13
  Metoprolol succinate | 3
  Metoprolol tartrate | 6
  Metronidazole | 1
  Milnacipran | 1
  Milnacipran hydrochloride | 1
  Mirtazapine | 4
  Mobizox | 1
  Molsidomine | 2
  Mometasone | 1
  Mometasone furoate | 1
  Montelukast | 3
  Montelukast sodium | 4
  Mosapride | 3
  Mosapride citrate | 7
  Moxifloxacin | 1
  Moxifloxacin hydrochloride | 3
  Mucaine | 1
  Multivitamins with minerals | 3
  Multivitamins, plain | 2
  Myprodol "rio ethicals" | 2
  Myrin plus | 1
  Myrtol | 3
  Naltrexone | 3
  Naproxen | 1
  Nateglinide | 4
  Nebivolol | 1
  Nicorandil | 5
  Nicotine | 3
  Nicotinic acid | 2
  Nifedipine | 16
  Nimesulide/paracetamol | 1
  Nimodipine | 2
  Nisoldipine | 1
  Nitrendipine | 1
  Nizatidine | 2
  Ofloxacin | 2
  Olanzapine | 2
  Olmesartan | 6
  Olmesartan medoxomil | 1
  Omega-3 marine triglycerides | 2
  Omega-3 triglycerides | 3
  Omeprazole | 9
  Ondansetron | 2
  Ondansetron hydrochloride | 1
  Orlistat | 4
  Oxazepam | 2
  Oxcarbazepine | 1
  Oxycodone | 1
  Oxycodone hydrochloride | 1
  Palonosetron hydrochloride | 1
  Pantoprazole | 7
  Pantoprazole sodium | 10
  Paracetamol | 9
  Paroxetine | 3
  Paroxetine hydrochloride | 3
  Pentamycin | 1
  Perindopril | 8
  Phenylephrine/triprolidine | 1
  Phenytoin sodium | 1
  Phosphatidyl choline | 1
  Phytomenadione | 1
  Pinaverium bromide | 1
  Pioglitazone | 4
  Pioglitazone hydrochloride | 4
  Platelets, human blood | 1
  Pneumococcal vaccine | 1
  Polycarbophil calcium | 2
  Pramipexole | 2
  Pranlukast hydrate | 1
  Pravastatin | 8
  Pravastatin sodium | 5
  Prednicarbate | 1
  Prednisolone | 5
  Pregabalin | 3
  Procaterol | 1
  Promethazine | 1
  Pronase | 2
  Propranolol | 2
  Propranolol hydrochloride | 2
  Propylthiouracil | 1
  Pseudoephedrine hydrochloride | 2
  Pyridostigmine bromide | 1
  Pyridoxine hydrochloride | 3
  Quetiapine fumarate | 2
  Rabeprazole | 9
  Rabeprazole sodium | 2
  Raloxifene | 1
  Ramipril | 7
  Ranitidine | 4
  Ranitidine hydrochloride | 3
  Rebamipide | 12
  Repaglinide | 3
  Rino ebastel | 1
  Riopan plus | 1
  Risedronic acid | 1
  Risperidone | 3
  Rosiglitazone maleate | 2
  Rosuvastatin | 24
  Rosuvastatin calcium | 1
  Roxithromycin | 2
  Salbutamol | 9
  Salbutamol sulfate | 1
  Salmeterol | 2
  Salmeterol xinafoate | 6
  Salvia miltiorrhiza | 1
  Sarpogrelate | 1
  Sarpogrelate hydrochloride | 2
  Selective beta-2-adrenoreceptor agonists | 1
  Selegiline hydrochloride | 1
  Seretide "allen & hanburys ltd" | 2
  Seretide mite | 17
  Sertraline | 2
  Sibutramine | 3
  Sibutramine hydrochloride | 1
  Sildenafil citrate | 2
  Silymarin | 2
  Simeco | 1
  Simvastatin | 21
  Sinemet | 1
  Sirolin retard | 2
  Sitagliptin | 6
  Sodium chloride | 1
  Sotalol hydrochloride | 1
  Spedifen | 1
  Spirapril hydrochloride | 1
  Spironolactone | 2
  Spironolactone / torasemide | 1
  Streptomycin | 1
  Sucralfate | 1
  Sulglicotide | 3
  Sulodexide | 1
  Symbicort turbuhaler "draco" | 11
  Tadalafil | 1
  Tamsulosin | 5
  Tamsulosin hydrochloride | 3
  Tazobactam sodium | 1
  Telmisartan | 17
  Terazosin | 1
  Terazosin hydrochloride | 1
  Terbinafine hydrochloride | 1
  Terbutaline | 3
  Terbutaline sulfate | 1
  Testosterone undecanoate | 1
  Theophylline | 18
  Thiamazole | 2
  Thioctic acid | 1
  Throat preparations | 1
  Tianeptine | 4
  Ticlopidine | 1
  Tiotropium | 10
  Tiotropium bromide | 3
  Tiotropium bromide/formoterol fumarate | 1
  Tiropramide hydrochloride | 3
  Tocopherol | 1
  Tolterodine | 1
  Tramadol | 1
  Tramadol hydrochloride | 1
  Tranexamic acid | 2
  Trazodone | 1
  Triaprin | 1
  Triazolam | 1
  Triflusal | 1
  Trihexyphenidyl | 1
  Trimebutine | 1
  Trimebutine maleate | 1
  Trimetazidine | 4
  Trimetazidine hydrochloride | 2
  Tromcardin | 1
  Udenafil | 2
  Ultracet | 3
  Ursodeoxycholic acid | 8
  Valproate semisodium | 1
  Valsartan | 10
  Varidase | 1
  Verapamil | 1
  Vildagliptin | 1
  Vitamin B | 1
  Vitamins | 1
  Vitamins with minerals | 1
  Vitamins, other combinations | 1
  Voglibose | 3
  Warfarin | 7
  Yeast | 1
  Zevit | 2
  Zinc | 1
  Zoledronic acid | 2
  Zolpidem | 10
  Zolpidem tartrate | 6

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Varenicline
Serious Adverse Events (participants affected / at risk) | 11/1373
Other Adverse Events (participants affected / at risk) | 379/1373
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=1373)
Acute myocardial infarction (Cardiac disorders) | 1
Cor pulmonale chronic (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Bronchiectasis (Infections and infestations) | 1
Haemorrhagic fever (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 1
Acute stress disorder (Psychiatric disorders) | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Varenicline (N=1373)
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Palpitations (Cardiac disorders) | 7
Hearing impaired (Ear and labyrinth disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal discomfort (Gastrointestinal disorders) | 11
Abdominal distension (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 3
Abdominal pain upper (Gastrointestinal disorders) | 12
Constipation (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 6
Dry mouth (Gastrointestinal disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 4
Epigastric discomfort (Gastrointestinal disorders) | 4
Eructation (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 1
Gastric disorder (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 8
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Hyperchlorhydria (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 156
Paraesthesia oral (Gastrointestinal disorders) | 1
Periodontitis (Gastrointestinal disorders) | 2
Regurgitation (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 12
Asthenia (General disorders) | 2
Chest discomfort (General disorders) | 3
Chest pain (General disorders) | 1
Fatigue (General disorders) | 11
Hunger (General disorders) | 1
Irritability (General disorders) | 3
Malaise (General disorders) | 2
Oedema peripheral (General disorders) | 1
Pyrexia (General disorders) | 1
Bronchitis (Infections and infestations) | 4
Gastroenteritis (Infections and infestations) | 2
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Nasopharyngitis (Infections and infestations) | 6
Otitis media chronic (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 2
Upper respiratory tract infection (Infections and infestations) | 7
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1
Drug exposure during pregnancy (Injury, poisoning and procedural complications) | 1
Fall (Injury, poisoning and procedural complications) | 1
Weight increased (Investigations) | 17
Decreased appetite (Metabolism and nutrition disorders) | 10
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Disturbance in attention (Nervous system disorders) | 2
Dizziness (Nervous system disorders) | 42
Dysgeusia (Nervous system disorders) | 7
Headache (Nervous system disorders) | 20
Hypersomnia (Nervous system disorders) | 2
Hypogeusia (Nervous system disorders) | 2
Lethargy (Nervous system disorders) | 2
Poor quality sleep (Nervous system disorders) | 3
Somnolence (Nervous system disorders) | 11
Abnormal dreams (Psychiatric disorders) | 28
Aggression (Psychiatric disorders) | 1
Agitation (Psychiatric disorders) | 2
Anxiety (Psychiatric disorders) | 7
Anxiety disorder (Psychiatric disorders) | 1
Bradyphrenia (Psychiatric disorders) | 4
Depression (Psychiatric disorders) | 4
Emotional disorder (Psychiatric disorders) | 1
Euphoric mood (Psychiatric disorders) | 1
Impatience (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 41
Listless (Psychiatric disorders) | 1
Restlessness (Psychiatric disorders) | 7
Sleep disorder (Psychiatric disorders) | 5
Albuminuria (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Renal pain (Renal and urinary disorders) | 1
Urinary hesitation (Renal and urinary disorders) | 1
Urinary tract disorder (Renal and urinary disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1
Menopausal symptoms (Reproductive system and breast disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sputum increased (Respiratory, thoracic and mediastinal disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 2
Essential hypertension (Vascular disorders) | 1
Hot flush (Vascular disorders) | 1
Hypertension (Vascular disorders) | 3

LIMITATIONS AND CAVEATS:
Outcome measures were not designated as primary or secondary measures as this study was a post-marketing, prospective, non-comparative and non-interventional study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.